CLINICAL TRIAL: NCT01232088
Title: Questionnaire of the Section Perioperative Intensive Care of the European Society of Intensive Care Medicine (ESICM) on Standardized Drug Labelling
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Department of Anesthesiology and Intensive Care Medicine CVK/CCM, Charite University, Berlin, Charite University, Berlin, Germany
Other Study IDs: Standardized Drug Labelling
Record Dates: First submitted 2010-11-01; First posted 2010-11-02 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Drug Labelling
Keywords: drug labelling; standardized drug syringe labelling; European ICU

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Data collection group: ICU physicians: Online survey for ICU physicians (members of the European Society of Intensive Care Medicine (ESICM)).

SUMMARY:
Medication errors are common in intensive care (Valentin A et al., BMJ. 2009;338). Standardized color coded labels for user applied syringes enjoy strong support from many health professionals, thinking that this might increase patient safety. Whether this is true or not warrants further research.

ELIGIBILITY:
Inclusion Criteria:

Members of the European Society of Intensive Care Medicine (ESICM)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Members of the European Society of Intensive Care Medicine (ESICM)
Sampling Method: Probability Sample
Enrollment: 482 (Actual)
Dates: Start 2010-11; Primary Completion 2011-06 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
The primary objective is to assess if standardized drug syringe labelling is used in European ICUs. | A period of 90 days.
  Online survey for ICU physicians (members of the ESICM).

SECONDARY OUTCOMES:
The second objectives is to assess 1. if standards for drug syringe labelling are similar in European ICUs and 2. if users expect that standardized drug syringe labelling should be delivered by the pharmaceutical industry. | A period of 90 days
  Online survey for ICU physicians (members of the ESICM).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine Campus Virchow Klinikum/Campus Charité Mitte, Berlin, State of Berlin, Germany

REFERENCES:
- [Background] Valentin A, Capuzzo M, Guidet B, Moreno R, Metnitz B, Bauer P, Metnitz P; Research Group on Quality Improvement of the European Society of Intensive Care Medicine (ESICM); Sentinel Events Evaluation (SEE) Study Investigators. Errors in administration of parenteral drugs in intensive care units: multinational prospective study. BMJ. 2009 Mar 12;338:b814. doi: 10.1136/bmj.b814. PMID 19282436
- [Derived] Balzer F, Wickboldt N, Spies C, Walder B, Goncerut J, Citerio G, Rhodes A, Kastrup M, Boemke W. Standardised drug labelling in intensive care: results of an international survey among ESICM members. Intensive Care Med. 2012 Aug;38(8):1298-305. doi: 10.1007/s00134-012-2569-1. Epub 2012 Apr 20. PMID 22527084